CLINICAL TRIAL: NCT00649753
Title: An Investigation of Algometer Readings for DeJarnette Category II Indicators After Category II Blocking and Cranial Protocol
Brief Title: Algometer and Category II Pelvic Blocking and Cranial Protocol
Acronym: Algometer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Mary Unger-Boyd, D.C., Logan College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SR0225080125
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2008-03

CONDITIONS: Pain; Sacroiliac Joint Dysfunction
Keywords: sacroiliac joint dysfunction; algometer; Chiropractic; Manual Therapy; indicator points associated with sacroiliac joint dysfunction
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- A (No Intervention)
- B (Experimental)
  Interventions: Procedure: Category II Pelvic Blocking
- C (Experimental)
  Interventions: Procedure: Category II Pelvic Blocking and Cranial
- D (Experimental)
  Interventions: Procedure: Cranial Only

INTERVENTIONS:
Procedure: Category II Pelvic Blocking — Supine Orthopedic Blocking consists of placing padded wedges underneath the Ilium and greater trochanter to correct pelvic torsion and associated sacroiliac dysfunction.
  Arms: B
Procedure: Category II Pelvic Blocking and Cranial — Supine Orthopedic Blocking consists of placing padded wedges underneath the Ilium and greater trochanter to correct pelvic torsion and associated sacroiliac dysfunction. During pelvic blocking a cranial procedure is performed using a zygomae release and sphenobasilar release. These cranial procedures are manual therapy procedures using light pressure from hand and/or finger contacts.
  Arms: C
Procedure: Cranial Only — Without pelvic blocking a cranial procedure is performed using a zygomae release and sphenobasilar release. These cranial procedures are manual therapy procedures using light pressure from hand and/or finger contacts.
  Arms: D

SUMMARY:
The purpose of this study is to evaluate the relationship of pelvic blocking and protocol for cranial adjusting with specific pain areas as outlined by Dr. Bertrand DeJarnette in the Category II/sacroiliac protocol. An algometer will be used to determine the level of pain at specific points before and after each treatment of pelvic blocking with or without cranial adjusting.

ELIGIBILITY:
Inclusion Criteria:

* Logan student, staff or faculty
* Age 18 - 60
* No chiropractic adjustment 2 weeks prior to beginning the study
* Show the DeJarnette Category II indicators

Exclusion Criteria:

* Previous lower extremity, first rib and spine injury, surgery
* Local infection, injury or other malignancy affecting the lower extremity and the nervous system
* Unstable joints of the lower extremity and/or first rib and/or spine
* Prescription or herbal muscle stimulants, relaxants, etc. that could affect the nervous system
* Contraindication to DeJarnette Category II Pelvis Blocking
* Pregnancy
* Significant lower lumbar involvement
* Diabetes, shortness of breath on light physical activity, cardiovascular disease
* Numbness and/or tingling in the lower extremities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Algometer readings | pre and post treatment intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Logan University, College of Chiropractic, Chesterfield, Missouri, United States